CLINICAL TRIAL: NCT02814214
Title: Device-based QRS Evaluation
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD_865
Record Dates: First submitted 2016-06-22; First posted 2016-06-27 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ECG+IEGM: Surface ECG and intracardiac electrogram recordings will be taken during the adjustment of programmable Cardiac Resynchronization Therapy settings
  Interventions: Device: ECG+IEGM

INTERVENTIONS:
Device: ECG+IEGM — Cardiac Resynchronization Therapy programming adjustments

SUMMARY:
The purpose of this study is to collect simultaneous surface electrocardiogram (ECG) recordings and Cardiac Resynchronization Therapy (CRT) intracardiac electrogram (IEGM) recordings of variations in electrical synchrony.

ELIGIBILITY:
Inclusion Criteria:

* Already implanted with SJM Quadripolar CRT Pacing System
* Ability to provide informed consent for study participation
* Willing to comply with the study evaluation requirements
* At least 18 years of age

Exclusion Criteria:

* Resting ventricular rate >100 bpm
* Intrinsic PR interval > 300 ms
* Paroxysmal or persistent atrial tachycardia or atrial fibrillation documented
* Pregnant or plans to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include approximately 100 patients who have been implanted with SJM Quadripolar Pacing Systems
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Characterize CRT IEGM-based estimations of QRS duration | Acute (1 day)

CONTACTS AND LOCATIONS:
Locations (1):
- I.R.C.C.S. Policlinico San Donato, San Donato Milanese, MI, Italy